CLINICAL TRIAL: NCT02222740
Title: A Multiple-Dose, Safety, Tolerability, and Pharmacokinetic Dose-Escalation Study of Hydrocodone Bitartrate Extended Release (HC-ER) in Patients With Chronic, Moderate to Severe Osteoarthritis Pain
Brief Title: A Safety, Tolerability and Pharmacokinetic Dose Escalation Study of HC-ER in Patients With Osteoarthritis Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ELN154088-203
Record Dates: First submitted 2014-07-21; First posted 2014-08-21 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2014-08

CONDITIONS: Osteoarthrosis
Keywords: Safety; Tolerability; Pharmacokinetics
MeSH Terms: conditions — Osteoarthritis | interventions — Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): 10 mg of Hydrocodone Bitartrate Extended Release (HC-ER) Twice per day (BID) for 7 days, followed by 20 mg BID for 7 days, followed by 30 mg BID for 7 days
  Interventions: Drug: 10 mg of Hydrocodone Bitartrate Extended Release (HC-ER)
- Group 2 (Experimental): 20 mg of Hydrocodone Bitartrate Extended Release (HC-ER) Twice Per Day (BID) for 7 days, followed by 30 mg BID for 7 days, followed by 40 mg BID for 7 days
  Interventions: Drug: 20 mg of Hydrocodone Bitartrate Extended Release (HC-ER)

INTERVENTIONS:
Drug: 10 mg of Hydrocodone Bitartrate Extended Release (HC-ER) — Schedule II Class
  Other Names: Zohydro ER
  Arms: Group 1
Drug: 20 mg of Hydrocodone Bitartrate Extended Release (HC-ER) — Schedule II Class
  Other Names: Zohydro ER
  Arms: Group 2

SUMMARY:
Assess the safety, tolerability and pharmacokinetics of multiple doses of 10, 20, 30, and 40 mg of Hydrocodone Bitartrate Extended Release (HC-ER)capsules taken with food at steady state, in subjects with chronic, moderate to severe osteoarthritis (OA) pain.

DETAILED DESCRIPTION:
Safety parameters assessed included adverse events, physical examinations, vital signs, 12-lead electrocardiogram (ECGs), clinical laboratory testing and overall Arthritis Pain Intensity and opioid side effects

ELIGIBILITY:
Inclusion Criteria:

* Subjects were 18 years or older
* Subjects had osteoarthritis (OA) defined by:

Presence of of typical hip and/or knee joint symptoms. Involvement of at least 1 hip or knee joints that had warranted treatment with Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), including cyclooxygenase-2 [COX-2] inhibitors and/or acetaminophen (APAP) for the last 3 months.

Radiographic evidence within the last 6 months of OA in the index joint, with Grade II to IV severity, as illustrated by the Atlas of Standard Radiographs.

* Subjects were otherwise in generally good health, as determined by the investigator, on the basis of medical history, physical examination, electrocardiogram (ECG), and screening laboratory results.
* Female subjects were either physically incapable of childbearing or were practicing an acceptable method of birth control and had a negative pregnancy test result demonstrated before dosing.
* Subjects had experienced a suboptimal response to APAP and NSAID therapy (including COX-2 inhibitor).
* Subjects had used opioids for OA pain on an as needed (PRN) or occasional basis.
* Subjects were willing and able to discontinue or modify their current medication used for management of OA pain per protocol.
* Subjects had steady, not transient, pain and a categorical pain rating of moderate to severe on a scale of none, mild, moderate, or severe.
* Subjects weighed > or = to100 lbs.
* If a subject had taken any inducers or inhibitors of cytochrome P450 [CYP450j), these were discontinued and an appropriate washout period (5 half-lives) had occurred before entry in the study.
* Subjects were able to take oral medication and were willing to comply with the protocol.
* Subjects agreed to abstain from alcohol consumption for the duration of the study.
* Subjects were able to read, understand, and voluntarily sign the IRB approved consent document before the performance of any study-specific procedures.

Exclusion Criteria:

* Subjects had any clinically significant condition that would, in the investigator's opinion, preclude study participation.
* Subjects had any other clinically significant form of disease at the index joint (study joint) or had been diagnosed with inflammatory arthritis, gout, pseudo-gout, Paget's disease, or any other chronic pain syndrome that, in the investigator's opinion, might interfere with the assessment of pain and other symptoms of OA.
* Subjects had known allergies or previous, significant reactions to opioids.
* Subjects had any laboratory abnormality at screening that was considered clinically significant by the investigator, or that, in the opinion of the investigator, would have contraindicated study participation.
* Subjects were known to have positive test results for human immunodeficiency virus (HIV), hepatitis B antigen, or hepatitis C antibody.
* Subjects had a history of chronic, scheduled opioid use for OA.
* Subjects had any signs or symptoms of opioid withdrawal.
* Subjects had a history of substance or alcohol abuse within 2 years before study entry.
* Subjects tested positively on a urine screen for drugs of abuse.
* Subjects had received any steroid therapy (e.g., oral, intramuscular, intravenous, or soft tissue) within 1 month of study entry.
* Subjects had a condition that would contraindicate the use of opioid analgesia.
* Subjects had participated in a study of an investigational drug or device, or had donated blood, within 30 days before study entry.
* Subjects used any medication that the investigator felt would interact unfavorably with the study medication (e.g., potentiation of sedation with tricyclic antidepressants).
* Subjects had used opioid analgesics for more than 3 days during the 30 days before screening.
* Subjects had a history of seizures.
* Subjects were considered by the investigator to be unsuitable for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2002-09; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Assess the steady-state pharmacokinetics (PK) of multiple dose of 10, 20, 30, and 40 mg of HC-ER | Day 1-28
  PK parameters including Tmax, Cmax and Cmin were calculated for each dose level in each group from the PK profile of hydrocodone and the metabolites hydromorphone, and norhydrocodone.